CLINICAL TRIAL: NCT02819973
Title: Educational Videos to Address Racial Disparities in Implantable Cardioverter Defibrillator Therapy Via Innovative Designs
Brief Title: Educational Videos to Address Racial Disparities in Implantable Cardioverter Defibrillator Therapy
Acronym: VIVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00071154
Record Dates: First submitted 2016-06-13; First posted 2016-06-30 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Sudden Cardiac Death; Heart Failure
Keywords: Patient Education; ICD; Implantable Cardioverter Defibrillator; Video; Decision; Decision making
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Educational Video 1 (Experimental): African American/ Black Video
  Interventions: Other: Educational Video1
- Educational Video 2 (Experimental): Caucasian Video
  Interventions: Other: Educational Video 2
- Usual Care (no video) 3 (Experimental): Standard Care/ No video
  Interventions: Other: Usual Care 3

INTERVENTIONS:
Other: Educational Video1
  Arms: Educational Video 1
Other: Educational Video 2
  Arms: Educational Video 2
Other: Usual Care 3
  Arms: Usual Care (no video) 3

SUMMARY:
VIVID is a prospective, multicenter, randomized clinical trial in African American patients that will to evaluate: (1) the effect of an educational video on knowledge of sudden cardiac death (SCD) and implantable cardioverter defibrillators (ICDs); (2) the effect of an educational video on the decision for ICD implantation, decisional conflict, and receipt of an ICD within 90 days; and 3) the effect of racial concordance between study patients and video participants (health care providers/patients) on the decision for ICD implantation, decisional conflict and ICD receipt within 90 days.

DETAILED DESCRIPTION:
VIVID is a prospective, multicenter, randomized clinical trial that will evaluate three specific research questions. In black patients eligible for a primary prevention implantable cardioverter defibrillator (ICD), 1) what is the effect of a patient-centered educational video compared with usual care (UC) on knowledge of SCD (Sudden Cardiac Death), associated risk factors, and ICDs; 2) what is the effect of a patient-centered educational video compared with UC on the decision for ICD implantation, decisional conflict, and receipt of an ICD within 90 days; 3) what is the effect of racial concordance between study patients and video participants (health care providers/patients) on the decision for ICD implantation, decisional conflict and ICD receipt within 90 days. In addition, in-depth qualitative interviews (IQI) with a sample of trial participants will be conducted to determine the salient influences on their decision and explore the reasons for their ultimate decision and subsequent implantation or non-implantation of an ICD.

Approximately 480 patients eligible for a primary prevention ICD will be enrolled at approximately 12 hospitals in this study. Study sites selected for VIVID will be geographically diverse and provide care to a significant proportion of racial and ethnic minority patients. Patient's will be mailed a letter regarding the study, prior to their initial visit. At the initial visit, patients will be approached about participation in the trial. For those interested, informed consent will be obtained and patients will be randomized. The investigators will be utilizing electronic consents on an iPad. Black patients will be randomized to one of 3 arms: educational videos presented in the same format; one with black participants (patients and providers) or the other with white participants (patients and providers); The third arm will be usual care (control) and the provider can interact with the patient consistent with their typical/usual care. Notably, for both intervention and control arms, all patient management decisions are completely at the discretion of the care providers.

ELIGIBILITY:
Inclusion Criteria:

1. Non-hospitalized patients with ejection fraction ≤35%
2. New York Heart Association class I-III heart failure,
3. Age >21
4. Eligible for an implantable cardioverter defibrillator (ICD) for the primary prevention of sudden cardiac death
5. Self-identified race as black
6. Provision of informed consent to participate in the study.

Exclusion Criteria:

1. Life expectancy <12 months
2. Listed for Orthotropic Heart Transplantation (OHT)
3. Transplant (OHT) or OHT imminent within 12 months,
4. History of ventricular fibrillation or sustained ventricular tachycardia without reversible causes
5. ICD already implanted
6. Myocardial infarction within the last 40 days,
7. Coronary revascularization within the last 3 months,
8. Patients who are unable to understand the study procedures due to cognitive or language barriers.
9. Inpatients will be excluded from the study because decision-making processes are thought to be appreciably different in inpatients as compared with outpatients.
10. Plan for subcutaneous ICD (Sub-Q ICD)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2016-07; Primary Completion 2020-01-28 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Thomas, MD, Principal Investigator — Duke University
Locations (14):
- United States (14):
  - University of California at San Francisco, San Francisco, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Arrhythmia Consultants and Research Institute, Macon, Georgia
  - Medstar Health Research Institute, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Jackson Heart, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - South Carolina Heart, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas KL, Al-Khatib SM, Kosinski AS, Sears SF Jr, Allen LaPointe NM, Jackson LR 2nd, Matlock DD, Haithcock D, Colley BJ 3rd, Hirsh DS, Peterson ED. Facilitating Shared Decision Making Among Black Patients at Risk for Sudden Cardiac Arrest : A Randomized Clinical Trial. Ann Intern Med. 2023 May;176(5):615-623. doi: 10.7326/M22-2934. Epub 2023 Apr 4. PMID 37011387
- [Derived] Thomas KL, Sullivan LT 2nd, Al-Khatib SM, LaPointe NA, Sears S, Kosinski AS, Jackson LR 2nd, Kutyifa V, Peterson ED. Videos to reduce racial disparities in ICD therapy Via Innovative Designs (VIVID) trial: Rational, design and methodology. Am Heart J. 2020 Feb;220:59-67. doi: 10.1016/j.ahj.2019.10.011. Epub 2019 Nov 11. PMID 31785550

RESULTS

PARTICIPANT FLOW:
Groups:
- Racially Concordant Video: Participants watching a video in which actors are primarily of the same race (Black/African American) as the participant
- Racially Discordant Video: Participants watching a video in which actors are primarily not of the same race (not Black/African American) as the participant.
- Usual Care (No Video): Standard Care/ No video
Period: Overall Study
Arm/Group | Racially Concordant Video | Racially Discordant Video | Usual Care (No Video)
Started | 114 | 114 | 115
Completed | 108 (2 withdrawn by request, 4 determined after randomization to be not eligible) | 111 (3 determined after randomization to be not eligible) | 111 (2 withdrawn by request, 2 determined after randomization to be not eligible)
Not Completed | 6 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Racially Concordant Video | Racially Discordant Video | Usual Care (no Video) | Total
Number analyzed (Participants) | 108 | 111 | 111 | 330
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.0 [52.3 to 68.7] | 59.0 [49.6 to 69.3] | 60.1 [53.8 to 68.8] | 59.3 [51.6 to 69.1]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 63 | 69 | 76 | 208
  Gender: Female | 44 | 42 | 35 | 121
  Gender: Unknown | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 108 | 111 | 111 | 330
Region of Enrollment [Number; unit: participants]
  United States | 108 | 111 | 111 | 330

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Saying "Yes" to ICD
Description: Proportion of patients who have decided by 7 days to receive an ICD among patients randomized to the video intervention compared with health care provider counseling (usual care)
Time Frame: 7 days
Population: Among patients randomized to the video intervention compared with health care provider counseling (usual care) and having outcome data recorded. Video arms were combined into a single group to measure the impact of video vs. no video.
Measure: Count of Participants; unit: Participants
Groups:
- Video: Participants randomized to watch a video about ICDs
- Usual Care (no Video): Participants randomized to usual care with no video
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 210 | 101
Participants
  Yes, want an ICD | 123 | 60
  No or unsure about an ICD | 87 | 41

2. Secondary Outcome: Proportion of Individuals Saying Yes to ICD Implant in the Racially Concordant Video
Description: Proportion of patients who watched a racially concordant video and who decided by 7 days to receive an ICD
Time Frame: 7 days
Population: All participants randomized to video arm for whom outcome data is available. Usual care arm is excluded from this outcome to measure the impact of racial concordance among those viewing a video.
Measure: Count of Participants; unit: Participants
Arm/Group | Racially Concordant Video | Racially Discordant Video
Number analyzed (Participants) | 102 | 108
Participants
  Yes, want an ICD | 54 | 69
  No or unsure about an ICD | 48 | 39

3. Secondary Outcome: Changes in Patient Knowledge (Pre and Post Intervention)
Description: Difference in Knowledge Questionnaire scores before and after receiving the intervention. Range of 0 to 13, with higher score indicating greater knowledge about ICDs.
Time Frame: Baseline preintervention and Baseline (approximately 20mins later) post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 218 | 111
score on a scale
  Pre-intervention knowledge score | 6.0 (2.6) | 6.1 (2.8)
  Post-intervention knowledge score | 9.0 (1.9) | 8.4 (2.4)

4. Secondary Outcome: Changes in Decisional Conflict (Pre and Post)
Description: Difference in Decisional Conflict Scale score from baseline pre-intervention to 1 week post-intervention, range of 0-100 with higher value indicating greater conflict about the decision to receive an ICD.
Time Frame: Baseline pre intervention and 1 week post intervention
Population: Among patients randomized to the video intervention compared with health care provider counseling (usual care) and having outcome data recorded at the specified time point. Video arms were combined into a single group to measure the impact of video vs. no video.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Usual Care (no Video): Participants randomized to receive usual care with no video
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 218 | 111
score on a scale
  Score baseline pre-intervention | 34.4 [25.0 to 44.9] | 37.5 [25.0 to 46.9]
  Score 1 week post-intervention: number analyzed (Participants) | 208 | 102
  Score 1 week post-intervention | 25.0 [12.5 to 28.1] | 25.0 [17.2 to 31.2]

5. Secondary Outcome: ICD Receipt Within 90 Days of Enrollment.
Description: Number of participants receiving ICD implant within 90 days of enrollment as assessed by medical record review.
Time Frame: 3 Months
Population: Among patients randomized to the video intervention compared with health care provider counseling (usual care) and having outcome data recorded at the specified timepoint. Video arms were combined into a single group to measure the impact of video vs. no video.
Measure: Count of Participants; unit: Participants
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 219 | 110
Participants | 142 | 74

6. Secondary Outcome: Time Spent With Patients by Providers in Each Arm of the Study
Description: Number of minutes spent with patients during baseline visit as measured by baseline questionnaire timer
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Video: Participants watching a video about ICDs.
- Usual Care (no Video): Participants not watching a video about ICDs.
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 201 | 110
minutes | 18.0 [9.0 to 31.0] | 20.0 [12.0 to 39.0]

7. Secondary Outcome: Patient Knowledge
Description: Assessment of knowledge retention at one week through re-administration of baseline Knowledge Questionnaire. Scale of 0-13, with higher score indicating more knowledge about ICDs.
Time Frame: 1 week
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Video | Usual Care (no Video)
Number analyzed (Participants) | 211 | 102
score on a scale | 9.0 [7.0 to 10.0] | 8.0 [6.0 to 10.0]

8. Other Pre Specified Outcome: In-depth Interview Focused on Barriers to ICD Placement Following the Initial Decision
Description: In-depth phone interview
Time Frame: 3 Month
Reporting Status: Not Posted

9. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Impact of the Video on the Decision
Description: In-depth phone interview
Time Frame: 3 Month
Reporting Status: Not Posted

10. Other Pre Specified Outcome: In-depth Interview Focused on Barriers to ICD Placement Following the Initial Decision
Description: In-depth phone interview
Time Frame: 1 week
Reporting Status: Not Posted

11. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Influences on the Decision to Accept or Decline an ICD
Description: In-depth phone interview
Time Frame: 3 Month
Reporting Status: Not Posted

12. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Impact of the Video on the Decision
Description: In-depth phone interview
Time Frame: 1 week
Reporting Status: Not Posted

13. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Knowledge of SCD and ICD
Description: In-depth phone interview
Time Frame: 3 Month
Reporting Status: Not Posted

14. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Influences on the Decision to Accept or Decline an ICD
Description: In-depth phone interview
Time Frame: 1 week
Reporting Status: Not Posted

15. Other Pre Specified Outcome: In-depth Qualitative Interviews Focused on Knowledge of SCD and ICD Therapy
Description: In-depth phone interview
Time Frame: 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: This was an intervention of a decision-making tool in standard care. Patients were followed for 90 days.
Description: This was an intervention of a decision-making tool in standard care. Death may have been reported spontaneously during attempts to contact a participant for a follow-up interview. No systematic efforts were made to collect adverse events, including mortality.
Groups:
- Educational Video 1: African American/ Black Video
  Educational Video1
- Educational Video 2: Caucasian Video
  Educational Video 2
- Usual Care (no Video) 3: Standard Care/ No video
  Usual Care 3
Arm/Group | Educational Video 1 | Educational Video 2 | Usual Care (no Video) 3
All-Cause Mortality (participants affected / at risk) | 0/108 | 4/111 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/111 | 0/111
Other Adverse Events (participants affected / at risk) | 0/108 | 0/111 | 0/111

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT02819973/SAP_000.pdf
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT02819973/Prot_001.pdf